CLINICAL TRIAL: NCT04246554
Title: Ketorolac as an Adjuvant Agent for Postoperative Pain Control Following Arthroscopic ACL Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospitals Cleveland Medical Center (Other)
Responsible Party: Principal Investigator, Michael Karns, MD., Principal Investigator, University Hospitals Cleveland Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: STUDY20180985
Record Dates: First submitted 2020-01-24; First posted 2020-01-29 (Actual); Results first posted 2021-12-21 (Actual); Last update posted 2021-12-21 (Actual); Status verified 2021-11

CONDITIONS: ACL Injury; Postoperative Pain
Keywords: ACL reconstruction; Ketorolac; Pain; Narcotic
MeSH Terms: conditions — Anterior Cruciate Ligament Injuries; Pain, Postoperative; Pain | interventions — Ketorolac; oxycodone-acetaminophen

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Control (Experimental): Patients receive oxycodone- acetaminophen (5mg-325mg) 28 tablets PRN for pain following ACL reconstruction surgery
  Interventions: Drug: Oxycodone-Acetaminophen
- Ketorolac (Experimental): Patients receive IV ketorolac followed by ketorolac 10 mg every 6 hours for 3 days following ACL reconstruction surgery. Patients are additionally discharged with oxycodone- acetaminophen (5mg-325mg) 28 tablets PRN for additional pain control
  Interventions: Drug: Ketorolac

INTERVENTIONS:
Drug: Ketorolac — Oral ketorolac for pain control following ACL reconstruction surgery
  Arms: Ketorolac
Drug: Oxycodone-Acetaminophen — Oral oxycodone-acetaminophen for post-operative pain control
  Arms: Control

SUMMARY:
1. The investigators aim to examine the use of IV and oral ketorolac as an adjunctive agent to the standard of care pain protocol for postoperative pain control following ACL reconstruction surgery.
2. The investigators hypothesize that the use of IV and oral ketorolac in addition to the standard of care pain protocol will reduce postoperative opioid consumption following ACL reconstruction surgery.

ELIGIBILITY:
Inclusion Criteria:

* Patients between 18 and 89 years old
* Patients undergoing primary anterior cruciate ligament (ACL) reconstruction surgery

Exclusion Criteria:

* Patients below age 18 or above age 89
* Illiterate or non-English speaking individuals
* Patients with contraindications to Ketorolac
* History of chronic alcohol or drug abuse
* Chronic use of psychotropic or analgesic drugs
* Known peptic ulcer disease or bleeding diasthesis
* Renal dysfunction (estimated glomerular filtration rate < 50 mL/min/1.73m2)
* Breastfeeding women
* Pregnant women

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 49 (Actual)
Dates: Start 2019-05-21 (Actual); Primary Completion 2020-10-09 (Actual); Study Completion 2021-01-01 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Michael Karns, MD, Principal Investigator — University Hospital Cleveland Medical Center
Locations (1):
- UH Cleveland Medical Center, Cleveland, Ohio, United States

REFERENCES:
- [Derived] Mengers SR, Strony JT, Sivasundaram L, Yu J, Goodfellow D, Salata MJ, Voos JE, Karns MR. Oral Ketorolac as an Adjuvant Agent for Postoperative Pain Control After Arthroscopic Anterior Cruciate Ligament Reconstruction: A Prospective, Randomized Controlled Study. J Am Acad Orthop Surg. 2022 Dec 15;30(24):e1580-e1590. doi: 10.5435/JAAOS-D-21-00721. PMID 36476466

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Control | Ketorolac
Started | 26 | 23
Completed | 26 | 22
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Control | Ketorolac | Total
Number analyzed (Participants) | 26 | 22 | 48
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 26 | 22 | 48
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 32.04 (12.98) | 31.91 (9.96) | 31.98 (11.57)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 17 | 12 | 29
  Male | 9 | 10 | 19
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 26 | 22 | 48
BMI [Mean (Standard Deviation); unit: kg/m^2] | 28.18 (6.19) | 28.03 (7.57) | 28.11 (6.80)
Smoker [Count of Participants; unit: Participants] | 5 | 3 | 8

OUTCOME MEASURES:

1. Primary Outcome: Postoperative Visual Analogue Scale Scores
Description: Patients will record their pain on a visual analogue scale with a minimum score of 0 and a maximum score of 100 where lower values indicate a lower pain level, and higher values indicate a higher pain level.
Time Frame: Up to 8 weeks postoperative
Measure: Mean (Standard Error); unit: score on a scale
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 26 | 23
score on a scale | 50.4 (5.3) | 40.0 (4.9)

2. Secondary Outcome: Narcotic Medication
Description: Number of oxycodone-acetaminophen tablets
Time Frame: 5 days
Measure: Mean (Standard Error); unit: tablets
Arm/Group | Control | Ketorolac
Number analyzed (Participants) | 26 | 23
tablets | 12.4 (1.4) | 5.5 (1.3)

ADVERSE EVENTS:
Time Frame: 6 weeks
Arm/Group | Control | Ketorolac
All-Cause Mortality (participants affected / at risk) | 0/26 | 0/22
Serious Adverse Events (participants affected / at risk) | 0/26 | 0/22
Other Adverse Events (participants affected / at risk) | 26/26 | 22/22
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Control (N=26) | Ketorolac (N=22)
nausea/ vomitin (Gastrointestinal disorders) | 5 (5) | 5 (5)
abdominal pain (Gastrointestinal disorders) | 1 (1) | 1 (1)
diarrhea (Gastrointestinal disorders) | 0 (0) | 0 (0)
constipation (Gastrointestinal disorders) | 3 (3) | 4 (4)
indigestion (Gastrointestinal disorders) | 0 (0) | 3 (3)
bleeding (Vascular disorders) | 0 (0) | 0 (0)
dizzy (Nervous system disorders) | 5 (5) | 2 (2)
drowsy (Nervous system disorders) | 11 (11) | 6 (6)
headache (Nervous system disorders) | 2 | 1 (1)

LIMITATIONS AND CAVEATS:
This is a single-institution study involving only five surgeons, so patient demographics and outcomes may not reflect a broader population. Neither surgeons nor patients were blinded with regards to medication use. Therefore, subjective pain scores may have been influenced by perceptions of greater pain control in patients who received ketorolac in addition to oxycodone-acetaminophen. The study may be underpowered with regards to functional outcome scores and medication side effects profiles.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (2):
  • Study Protocol and Statistical Analysis Plan (2019-05-09): https://cdn.clinicaltrials.gov/large-docs/54/NCT04246554/Prot_SAP_000.pdf
  • Informed Consent Form (2019-05-21): https://cdn.clinicaltrials.gov/large-docs/54/NCT04246554/ICF_001.pdf